CLINICAL TRIAL: NCT04159389
Title: Learning Mental Visualization to Improve Performance in Anesthesia: a Randomized Controlled Trial by Simulation
Brief Title: Mental Visualization as a Learning Tool in Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Grenoble Alps (Other)
Responsible Party: Principal Investigator, Pierre ALBALADEJO, Clinical Professor, University Grenoble Alps
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CESAR002
Record Dates: First submitted 2019-10-26; First posted 2019-11-12 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Anesthesia; Medical Education
Keywords: airway management; pedagogy; learning process; mental visualization; rapide sequence induction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional teaching (No Intervention): theoretical courses and procedural simulation on airway management during rapid sequence induction
- Mental visualization (Experimental): traditional teaching completed by mental visualization : theoretical courses and procedural simulation on airway management during rapid sequence induction + mental visualization (theoretical courses, audioguide for individual practice and experience sharing session)
  Interventions: Other: Mental visualization

INTERVENTIONS:
Other: Mental visualization — Instruction in mental visualization by theoretical lessons and support of practice by audio guide and session of experience sharing.
  Arms: Mental visualization

SUMMARY:
The purpose of this study is to evaluate the benefit of adding mental visualization to a training program in medical education. Undergraduate medical students will be randomized before participating in a training program on airway management during rapid sequence induction. In the control group, participants will receive traditional teaching including theoretical courses and procedural simulation. In the intervention group, in addition to traditional teaching, participants will be trained and encouraged to practice mental visualization. The main outcome will be clinical performance during a standardized high-fidelity simulation of rapid sequence induction assessed using a specific pre-established checklist.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate medical students from the Grenoble Alps university hospital
* From the 2nd to the 6th year
* Volontary

Exclusion Criteria:

* /

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2022-03-05 (Actual)

PRIMARY OUTCOMES:
Clinical performance for airway management in a standardized high-fidelity simulation of rapid sequence induction. | 2 weeks
  All simulations will be videotaped and the clinical performance of each participant will be assessed by an independent evaluator using a specific pre-established checklist

SECONDARY OUTCOMES:
"Material preparation" score, subpart 1 of the clinical performance grid | 2 weeks
  All simulations will be videotaped and the score of the subpart "Material preparation" of the clinical performance of each participant will be assessed by an independent evaluator using a specific pre-established checklist
"Intubation procedure" score, subpart 2 of the clinical performance grid | 2 weeks
  All simulations will be videotaped and the score of the subpart "Intubation procedure" of the clinical performance of each participant will be assessed by an independent evaluator using a specific pre-established checklist
Physiological stress response : SDNN | 2 weeks
  Heart rate variability evaluated by SDNN (Standard Deviation Normal to Normal), in miliseconds. Physiological stress response is higher when SDNN is lower.
Psychological stress response : Stress-VAS | 2 weeks
  Stress Visual Analogical Scale, from 0 to 100, psychological stress response is higher when score is higher.
Psychological stress response : STAI | 2 weeks
  STAI (State-Trait Anxiety Inventory), from 20 to 80, psychological stress response is higher when score is higher.
Adesion to Mental visualization | 2 weeks
  Frequency questionnaire for the use of mental visualization, from "0" to ">1 per day". We ask the participant to use it once a day
Quality to Mental visualization : MIQ | 2 weeks
  Mental Imagery Questionnaire, from 8 to 56, mental visualisation is better when score is higher.
Memorization of key messages at three months | 3 months
  Specific pre-established checklist : 5-point grid. Assessed by an independent evaluator using a phone call.

CONTACTS AND LOCATIONS:
Locations (1):
- University Grenoble Alps, La Tronche, France

IPD SHARING:
Plan to Share IPD: Undecided